CLINICAL TRIAL: NCT01407952
Title: New Generation Hydrogel Endovascular Aneurysm Treatment Trial
Brief Title: Hydrogel Endovascular Aneurysm Treatment Trial
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: MicroVention, Inc. (Industry)
Responsible Party: Principal Investigator, Bernard Bendok, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEAT_protocol1
Record Dates: First submitted 2011-07-12; First posted 2011-08-02 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Aneurysm
Keywords: treatment trial; cerebral aneurysm; randomized; coils; endovascular; HEAT; bare platinum; Hydrogel; Hydrocoil
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HydroCoil Embolic System (Other): Aneurysm treatment using the HydroCoil Embolization System (21 CFR 882.5950)
  Interventions: Device: HydroCoil Embolic System
- Control (Other): Aneurysm treatment using bare platinum coil(s)
  Interventions: Device: Control (bare platinum coils)

INTERVENTIONS:
Device: HydroCoil Embolic System — HydroCoil Embolic System
  Other Names: MicroVention, Inc
  Arms: HydroCoil Embolic System
Device: Control (bare platinum coils) — bare platinum coils
  Arms: Control

SUMMARY:
This research study is being done to test the effectiveness of a new generation FDA approved device for treating aneurysms compared to the current standard device for endovascular aneurysm treatment which is bare platinum coils. Endovascular procedures are a form of minimally invasive surgery, which is performed on blood vessels. The technique involves the introduction of a catheter which is a long, thin, flexible, hollow plastic tube through the skin into a large blood vessel. Typically the chosen blood vessel is the femoral artery found near the groin. The catheter is then maneuvered through the body to the location of the aneurysm in the brain using image guidance. Coils are delivered into the aneurysm through the catheters. Once the coils are delivered in the aneurysm, they are detached from the catheter. This is repeated until enough coils fill the aneurysm, blocking the blood flow to the aneurysm. The body responds by forming blood clots around the coil(s), which helps block the flow of blood into the aneurysm and keeps the vessel from rupturing or leaking. This study will compare the study device to the standard bare platinum coil to see which is better at preventing future rupturing or leaking. The study device is called the HydroCoil Embolization System and this study is a post-market clinical trial.

About 600 subjects from multiple institutions will take part in this study.

DETAILED DESCRIPTION:
Your part in this study will last up to 24 months and will involve 6 visits (1 baseline visit before your surgery, the surgical procedure and 4 follow-up visits). These visits will occur at the same time as the visits you would receive as standard of care after your surgery.

If you are in this study, you will be placed in one of two study groups by chance using a process similar to the flip of a coin. This process is called randomization. Neither you nor the study staff will select the group you will be in. One group, the control group, will have their aneurysm treated by the bare platinum coils during their endovascular procedure. The other group, the study group will receive coils from the HydroCoil Embolization System. Both groups will receive the same standard of care and follow-up, but during the surgery different types of coils will be used.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet the following criteria to be enrolled in the study:

1. Patient is between 18 and 75 years of age (inclusive).
2. Patient has a documented untreated intracranial saccular aneurysm 3-14 mm diameter angiographic lumen, ruptured or unruptured, suitable for embolization with coils.
3. Patients presenting with a HUNT and HESS Grade 0-3 or improving to such a grade before treatment
4. Any type of bare platinum coils and HydroCoil ® Coils are treatment options (all shapes allowed).
5. Patient or next of kin or person with appropriate power of attorney has provided written informed consent.
6. Patient is willing and available for study follow-up visits
7. Patient has not been previously entered into this Study

Exclusion Criteria:

Candidates will be ineligible for enrollment in the study if any of the following conditions apply:

1. Inability to obtain informed consent
2. Patient is < 18 or > 75 years old
3. Target aneurysm is not saccular in nature (mycotic, fusiform, dissecting).
4. Target aneurysm is > 14 mm maximum luminal dimension, < 3 mm maximum luminal dimension
5. Target aneurysm has been previously clipped or coiled
6. Target aneurysm is in the physician's estimate unlikely to be successfully treated by endovascular techniques.
7. Patient has known hypersensitivity to platinum, nickel, stainless steel or structurally related compounds found in HydroCoil®, HydroSoft®, HydroFrame® Coils and/or bare platinum coils.
8. Baseline Hunt and Hess scale 4 or 5 for ruptured aneurysms
9. Intended use of a flow diverting stent (e.g. pipeline)
10. Subject has concurrent intracranial pathology, e.g.

    * Moyamoya
    * Vasculitis documented by biopsy results
    * AVMs
    * AV fistulas
    * Significant atherosclerotic disease (i.e. symptomatic and or >50% narrowing of the parent arteries necessary to traverse in order to coil the target aneurysm)
    * Intracranial Hematoma (unrelated to the target aneurysm)
    * Brain tumors
    * Vascular tortuosity and other conditions preventing access to target aneurysm
11. Subject has serious co-morbidities that could confound the study results:

    * Uncontrolled hypertension
    * Uncorrectable coagulation abnormality
    * Contraindications for heparin, aspirin or clopidogrel
    * Uncontrolled Diabetes Mellitus
    * Organ failure of kidney, liver, heart, or lung
    * Myocardial infarction within the past 6 months
    * Cancer likely to cause death within 2 years or less.
12. Subject history indicates high risk of non-compliance (e.g., substance abuse, psychosocial issues, etc.)
13. Subject has a known history contraindicating contrast dye or iodine that cannot be pre-medicated prior to coiling procedure (vs. sensitivity which can be safely controlled by antihistamine, steroid, etc.). Medical clearance will be needed for this issue.
14. Patients who are unable to complete scheduled follow up assessments at the enrolling center due to limited life expectancy (<2 years), co-morbidities or geographical considerations
15. Subject is currently breast feeding, pregnant or plans to become pregnant in the next 2 years.
16. Major surgical procedure or trauma within 30 days prior to randomization
17. The patient is currently enrolled in another clinical study (device or drug).
18. More than one aneurysm needing treatment at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard R Bendok, MD, Principal Investigator — Mayo Clinic
Locations (44):
- United States (38):
  - St. Joseph's Hospital, Phoenix, Arizona
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Christiana Hospital, Newark, Delaware
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Queens Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Advocate Health, Oak Lawn, Illinois
  - University of Louisville, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Consulting Radiologists, LTD, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - SUNY Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Kaiser Permanente NW, Clackamas, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hamot, Erie, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Hospital Research Institute, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - MultiCare Health System, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (6):
  - Dalhousie Univerisity, Halifax, Nova Scotia
  - Hamilton Health/McMaster Univeristy, Hamilton, Ontario
  - CHUM Research Centre, Montreal, Quebec
  - McGill Universtiy, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
  - CHU de Quebec, Québec

REFERENCES:
- [Derived] Bendok BR, Abi-Aad KR, Ward JD, Kniss JF, Kwasny MJ, Rahme RJ, Aoun SG, El Ahmadieh TY, El Tecle NE, Zammar SG, Aoun RJN, Patra DP, Ansari SA, Raymond J, Woo HH, Fiorella D, Dabus G, Milot G, Delgado Almandoz JE, Scott JA, DeNardo AJ, Dashti SR; HEAT Study Investigators. The Hydrogel Endovascular Aneurysm Treatment Trial (HEAT): A Randomized Controlled Trial of the Second-Generation Hydrogel Coil. Neurosurgery. 2020 May 1;86(5):615-624. doi: 10.1093/neuros/nyaa006. PMID 32078692

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HydroCoil Embolic System | Control
Started | 297 | 303
Completed | 251 | 266
Not Completed | 46 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HydroCoil Embolic System | Control | Total
Number analyzed (Participants) | 297 | 303 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.5) | 56.9 (10.3) | 56.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 236 | 474
  Male | 59 | 67 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 243 | 247 | 490
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 32 | 27 | 59
  White | 243 | 247 | 490
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Aneurysm Recurrence Post Surgery
Description: Defined as any progression on the Raymond-Roy (RR) Aneurysm Occlusion Scale. The RR scale is such that 1=complete occlusion, 2=residual neck, and 3=residual aneurysm.
Time Frame: post surgery to 24 months
Measure: Number; unit: participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 251 | 266
participants | 11 | 41
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; A intent to treat analysis was performed, using multiple imputation methods; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.36 to 3.97]
Statistical Analysis 2: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p < 0.01, Chi-squared — Chi-squared test statistic with one degree of freedom=17.37; Odds Ratio (OR) = 3.97, 95% CI 2-sided [1.99 to 7.92]

2. Secondary Outcome: Packing Density
Description: Packing density as measured by volumetric filling of the aneurysm
Time Frame: at operation
Population: Participants with both imaging data (to determine aneurysm size), and coil information (length, number, and type used)
Measure: Mean (Standard Deviation); unit: density as expressed as a percentage
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 238 | 237
density as expressed as a percentage | 32.5 (14.8) | 24.7 (10.2)
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Clinical Outcome: Modified Rankin Scale (mRS)
Description: modified rankin scale is a measure of neurological disability, which ranges from 0=no symptoms to 5=severe disability (6=dead).
Time Frame: 24 months
Population: Based on participants with any post procedural follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 287 | 292
Participants
  No symptoms (mRS=0) | 181 | 178
  No significant disability (mRS=1) | 60 | 63
  Slight disability (mRS=2) | 24 | 28
  Moderate disability (mRS=3) | 13 | 10
  Moderately severe disability (mRS=4) | 2 | 0
  Severe disability (mRS=5) | 0 | 4
  Expired (mRS=6) | 7 | 9
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.578, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Adverse Events Related to the Procedure and/or the Device by Participant at Any Time in the Study.
Description: number of participants who experienced any peri-procedural or post-procedural Adverse Event noted to be related to the procedure or device.
Time Frame: 24 months
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 297 | 303
Participants | 64 | 75
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.352, Chi-squared; Chi-squared test statistic with one degree of freedom = 0.865

5. Secondary Outcome: Total Number of Peri-procedural and Post-procedural Adverse Events Related to the Procedure and/or the Device.
Description: total number of Adverse Events per person that were noted to be related to the procedure and device during the study
Time Frame: 24 months
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 297 | 303
Participants
  No events | 233 | 228
  One event | 44 | 63
  Two events | 19 | 8
  Three events | 1 | 4
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.769, Cochran-Armitage Trend Test

6. Secondary Outcome: Number of Patients Who Expired During the Study (Mortality Rate)
Description: all-cause mortality at any time during study follow-up
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 297 | 303
Participants | 7 | 9
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.641, Chi-squared; Chi-square test statistic with one degree of freedom=0.217

7. Secondary Outcome: Number of Participants With Initial Complete Occlusion
Description: Raymond-Roy (RR) Scale=1 at procedure The RR scale is such that 1=complete occlusion, 2=residual neck, and 3=residual aneurysm.
Time Frame: at procedure
Population: Raymond-Roy Scale recorded at procedure
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 281 | 290
Participants | 50 | 82
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.003, Chi-squared; chi-square test statistic with one degree of freedom=8.82

8. Secondary Outcome: Number of Patients Who Needed Re-treatment of Target Aneurysm
Description: During the 24 month follow-up, if Aneurysm needed to be re-treated.
Time Frame: 24 months
Population: participants with available followup
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 251 | 266
Participants | 13 | 22
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.162, Chi-squared; Chi-squared test statistic with one degree of freedom=1.955

9. Secondary Outcome: Number of Participants Experiencing a Hemorrhage From Target Aneurysm Post Surgery
Description: Per the Adverse event log, if a hemorrhage or rupture occurred that was noted to be related to the procedure or device at any point during the 24 month follow-up (not during the operation).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 297 | 303
Participants | 2 | 0
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p = 0.245, Fisher Exact

10. Secondary Outcome: Number of Participants Who Progressed on the Meyers Scale
Description: Occlusion (in)stability was determined by progression on the Meyers scale. The Meyer scale is a 6-point grading scale based on the percentage of the aneurysm filled by contrast on DSA. Grade zero indicates complete and total aneurysm occlusion without remnant or in-terstitial filling within the aneurysm. Grade 1 represents greater than 90%volumetric occlusion of the aneurysm based on planar imaging assessment; grade 2, 70%-89% aneurysm occlusion; grade 3,50%-69%; grade 4, 25%-49%; and grade 5, less than 25% volumetric aneurysm occlusion.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 251 | 266
Participants | 33 | 71
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p < 0.01, Chi-squared; Chi-squared test statistic with one degree of freedom=14.743

11. Secondary Outcome: Number of Participants Experiencing Major Versus Minor Recurrence by 24 Months Follow-up.
Description: Major recurrence is defined as progression on the Raymond-Roy (RR) Scale to 3, or if initial RR was 3, then progression on the Meyers scale. Minor recurrence was defined as a progression on the RR scale to 2.
  The RR scale is a 3 point measure of occlusion, 1=total, 2=residual neck, and 3=residual aneurysm.
  The Meyer scale is a 6-point grading scale based on the percentageof the aneurysm filled by contrast on DSA. Grade zero indicates complete and total aneurysm occlusion without remnant or in-terstitial filling within the aneurysm. Grade 1 represents >90%volumetric occlusion of the aneurysm based on planar imaging assessment; grade 2, 70%-89% aneurysm occlusion; grade 3,50%-69%; grade 4, 25%-49%; and grade 5, <25% volumetric aneurysm occlusion.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | HydroCoil Embolic System | Control
Number analyzed (Participants) | 251 | 266
Participants
  Major recurrence | 32 | 55
  Minor recurrence | 2 | 14
  No major/minor recurrence | 217 | 197
Statistical Analysis 1: Comparison: HydroCoil Embolic System vs Control; Test type: Superiority; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data was collected until 18-24 month visit.
Arm/Group | HydroCoil Embolic System | Control
All-Cause Mortality (participants affected / at risk) | 7/297 | 9/303
Serious Adverse Events (participants affected / at risk) | 61/297 | 69/303
Other Adverse Events (participants affected / at risk) | 118/297 | 140/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HydroCoil Embolic System (N=297) | Control (N=303)
Air embolism (Surgical and medical procedures) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Aneurysm, left ICA ophthalmic (Nervous system disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Arrythmia (Cardiac disorders) | 1 (1) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy, non-schemic (Cardiac disorders) | 1 (1) | 1 (1)
Carotid artery dissection (Vascular disorders) | 0 (0) | 2 (2)
Cerebral salt wasting (Renal and urinary disorders) | 0 (0) | 1 (1)
Coil herniation (Surgical and medical procedures) | 1 (1) | 0 (0)
Coil prolapse (Surgical and medical procedures) | 1 (1) | 1 (1)
Concussion (Nervous system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture left-femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin hematoma (Surgical and medical procedures) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 5 (5)
Hemianopsia (Eye disorders) | 0 (0) | 2 (2)
Hemorrhage, intraventicular (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 8 (9) | 4 (4)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Intracranial aneurysm, ruptured (Nervous system disorders) | 3 (3) | 6 (6)
Intracranial hemorrhage, non-specified (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage, subarachnoid (Nervous system disorders) | 2 (2) | 1 (1)
Intracranial, hemorrhage, subdural (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Leukocytosis (Infections and infestations) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 2 (2)
Parasthesia (Nervous system disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Psedudoaneurysm, cerebral (Vascular disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Retroperitonial hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Scotoma (Eye disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 7 (9) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 15 (16) | 11 (11)
Transient ischemic attach (Nervous system disorders) | 0 (0) | 1 (1)
Procedural Thrombosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 11 (16) | 17 (19)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HydroCoil Embolic System (N=297) | Control (N=303)
Headache (Nervous system disorders) | 38 (49) | 50 (53)
Vasospasm (Vascular disorders) | 15 (15) | 18 (18)
Visual Disturbance (Eye disorders) | 17 (17) | 30 (31)
Parasthesia (Nervous system disorders) | 8 (9) | 14 (14) — Numbness in face, arms, legs
Other (General disorders) | 70 (105) | 86 (111) — All other adverse events that did not meet the 3% threshold individually. (e.g. Anemia, Dyspnea, Rash)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT01407952/Prot_SAP_000.pdf